CLINICAL TRIAL: NCT00817635
Title: A Phase II, Randomized, Double-blind, Placebo and Active Controlled, Parallel Group, Multi-center, Dose Ranging Study to Evaluate the Efficacy and Safety of LCI699 Compared to Placebo After 8 Weeks Treatment in Patients With Resistant Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of LCI699 Compared to Placebo in Participants With Resistant Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Great Lakes Drug Development, Inc. (Industry); Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCI699A2216; 2008-007338-23 (EudraCT Number)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Blood Pressure; Hypertension; Resistant Hypertension
MeSH Terms: conditions — Hypertension | interventions — Osilodrostat; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LCI699 0.25 mg BID (Experimental): Following a 2-week placebo run-in period, participants received LCI699 0.25 mg, capsules, orally, twice daily (BID), with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- LCI699 1 mg QD (Experimental): Following a 2-week placebo run-in period, participants received LCI699 1 mg, capsules, orally, once daily (QD), with or without food for up to 8 weeks.
  Interventions: Drug: LCI699
- LCI699 0.5 mg followed by LCI699 1 mg BID (Experimental): Following a 2-week placebo run-in period, participants received LCI699 0.5 mg, capsules, orally, BID, with or without food for up to 4 weeks, followed by LCI699 1 mg, capsules, orally, BID with or without food for up to 4 weeks.
  Interventions: Drug: LCI699
- Eplerenone 50 mg BID (Active Comparator): Following a 2-week placebo run-in period, participants received eplerenone 50 mg, capsules, orally, BID, with or without food for up to 8 weeks.
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator): For a 2-week placebo run-in period, followed by 8 weeks of the treatment period, participants received LCI699-matching placebo or eplerenone-matching placebo, capsules, orally, QD or BID, with or without food.
  Interventions: Drug: LCI699-matching Placebo; Drug: Eplerenone-matching Placebo

INTERVENTIONS:
Drug: LCI699 — LCI699 oral capsules
  Arms: LCI699 0.25 mg BID; LCI699 0.5 mg followed by LCI699 1 mg BID; LCI699 1 mg QD
Drug: Eplerenone — Eplerenone oral capsules
  Arms: Eplerenone 50 mg BID
Drug: LCI699-matching Placebo — LCI699-matching placebo oral capsules
  Arms: Placebo
Drug: Eplerenone-matching Placebo — Eplerenone-matching placebo oral capsules
  Arms: Placebo

SUMMARY:
This study assessed the blood pressure effect, safety and tolerability of LCI699 compared to placebo and eplerenone in participants with resistant hypertension.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of hypertension with mean sitting systolic blood pressure (MSSBP) ≥140 millimeters of mercury (mmHg) and <180 mmHg
* Stable on a three-drug regimen (including a diuretic) for at least 4 weeks for the treatment of resistant hypertension
* Male and female participants 18 to 75 years of age

Exclusion criteria:

* Recent history of myocardial infarction (MI), heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack
* Clinically significant electrocardiography (ECG) findings related to cardiac conduction defects
* Type 1 diabetes or uncontrolled type 2 diabetes (haemoglobin A1c [HbA1c] >9%)
* Malignancies within the last 5 years (excluding basal cell skin cancer)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2008-12-22 (Actual); Primary Completion 2009-10-13 (Actual); Study Completion 2009-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (37):
  - Horizon Research Group, Inc, Mobile, Alabama
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Clinical Solutions Advantage, Buena Park, California
  - Michael Waldman, MD, Irvine, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Clinical Trials Research, Roseville, California
  - Orange County Research Center, Tustin, California
  - Metro Clinical Research, Littleton, Colorado
  - Meridien Research, Bradenton, Florida
  - Clinical Research of So. Florida, Coral Gables, Florida
  - Jacksonville Heart Center, Jacksonville Beach, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Accelovance, Melbourne, Florida
  - Cardio-Pulminary Associates, Plantation, Florida
  - Meridien Research, St. Petersburg, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Provident Clinical Research, Addison, Illinois
  - Cedar-Crosse Research Centereet, Chicago, Illinois
  - Provident Clinical Research, Bloomington, Indiana
  - Accelovance, South Bend, Indiana
  - Peter A. Holt, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Chelsea Internal Medicine, Chelsea, Michigan
  - New York Cardiovascular Associates, New York, New York
  - Charlotte Clinical Research, Charlotte, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Community Research, Cincinnati, Ohio
  - Tipton Medical & Diagnostic Center, Tipton, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - Mountain View Clinical Research Associates, Greer, South Carolina
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Punzi Medical Center, Carrollton, Texas
  - KRK Medical Research, Dallas, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Daniel Gottlieb, MD, Burien, Washington
  - Rainier Clinical Research Center, Renton, Washington
  - Gemini Scientific, Madison, Wisconsin
- Encode Clinic, Reykjavik, SA, Iceland

REFERENCES:
- [Derived] Schumacher CD, Steele RE, Brunner HR. Aldosterone synthase inhibition for the treatment of hypertension and the derived mechanistic requirements for a new therapeutic strategy. J Hypertens. 2013 Oct;31(10):2085-93. doi: 10.1097/HJH.0b013e328363570c. PMID 24107737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 35 investigative sites in the United States and in Iceland from 22 December 2008 to 13 October 2009.
Pre-assignment Details: Participants with a diagnosis of resistant hypertension were enrolled in a run-in period (Week -2 to 0). After that, the participants who fulfilled the inclusion criteria and did not meet any of the exclusion criteria at Week -2 and Week 0 were randomized to receive LCI699 or eplerenone in comparison with placebo for 8 weeks.
Period: Overall Study
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Started | 32 | 26 | 31 | 33 | 33
Completed | 23 | 22 | 28 | 28 | 25
Not Completed | 9 | 4 | 3 | 5 | 8
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1
Not completed — Abnormal Laboratory Value(s) | 1 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Administrative Problems | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 5 | 1 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) population included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo | Total
Number analyzed (Participants) | 32 | 26 | 31 | 33 | 33 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (10.36) | 55.4 (9.58) | 57.2 (10.77) | 56.2 (7.70) | 59.8 (9.33) | 56.5 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 13 | 14 | 11 | 58
  Male | 20 | 18 | 18 | 19 | 22 | 97
Baseline Mean Sitting Systolic Blood Pressure (MSSBP) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] | 152.4 (11.21) | 152.5 (9.79) | 152.2 (7.58) | 153.8 (8.92) | 153.4 (9.61) | 152.9 (9.39)
Baseline Mean Sitting Diastolic Blood Pressure (MSDBP) [Mean (Standard Deviation); unit: mmHg] | 91.8 (11.68) | 89.2 (9.56) | 88.9 (11.89) | 89.1 (9.84) | 90.1 (11.65) | 89.8 (10.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MSSBP at Week 8 Last Observation Carried Forward (LOCF)
Description: Arterial blood pressure (BP) determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in the MSSBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from Baseline in MSSBP was analyzed using an analysis of covariance model (ANCOVA) with treatment and country as factors and Baseline MSSBP as a covariate.
Time Frame: Baseline, Week 8
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug. Overall number of participants analyzed signifies the number of participants who were evaluable for this measure.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
mmHg | -11.4 (2.96) | -13.1 (3.24) | -12.5 (2.96) | -18.7 (2.92) | -8.8 (2.87)

2. Secondary Outcome: Change From Baseline in MSDBP at Week 8 LOCF
Description: Arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in the MSDBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from Baseline in MSDBP was analyzed using an ANCOVA with treatment and country as factors and Baseline MSDBP as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
mmHg | -4.5 (1.72) | -6.0 (1.88) | -6.1 (1.72) | -7.7 (1.69) | -4.8 (1.66)

3. Secondary Outcome: Percentage of Participants With a MSSBP Response and MSSBP Control at Week 8, as Measured by Office Blood Pressure (OBP)
Description: MSSBP response was defined as the percentage of participants with a MSSBP <140 mmHg or a >=20 mmHg reduction from baseline reduction from baseline. MSSBP control was defined as the percentage of participants with a MSSBP <140 mmHg for non-diabetic participants and <130mHg for diabetic participants.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- LCI699 0.25 mg BID: Following a 2-week placebo run-in period, participants received LCI699 0.25 mg capsules, orally, twice daily (BID), with or without food for up to 8 weeks.
- LCI699 1 mg QD: Following a 2-week placebo run-in period, participants received LCI699 1 mg capsules, orally, once daily (QD), with or without food for up to 8 weeks.
- LCI699 0.5 mg Followed by LCI699 1 mg BID: Following a 2-week placebo run-in period, participants received LCI699 0.5 mg capsules, orally, BID, with or without food for up to 4 weeks, followed by LCI699 1 mg capsules, orally, BID, with or without food for up to 4 weeks.
- Eplerenone 50 mg BID: Following a 2-week placebo run-in period, participants received eplerenone 50 mg capsules, orally, BID, with or without food for up to 8 weeks.
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
percentage of participants
  MSSBP Response | 54.8 | 57.7 | 41.9 | 65.6 | 42.4
  MSSBP Control | 51.6 | 50.0 | 32.3 | 53.1 | 36.4

4. Secondary Outcome: Percentage of Participants With a MSDBP Response and MSDBP Control at Week 8, as Measured by OBP
Description: MSDBP response was defined as the percentage of participants with a MSDBP <90 mmHg or a >=10 mmHg reduction from baseline. MSDBP control was defined as the percentage of participants with a MSDBP <90 mmHg for non-diabetic participants and <80mHg for diabetic participants.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
percentage of participants
  MSDBP Response | 67.7 | 73.1 | 71.0 | 71.9 | 57.6
  MSDBP Control | 54.8 | 65.4 | 58.1 | 56.3 | 54.5

5. Secondary Outcome: Dose/Exposure BP Response Relationship of LCI699, as Measured by Change From Baseline in MSSBP at Week 8
Description: Arterial BP determinations were made after the participant was in the sitting position for 5 minutes according to the American Heart Association guidelines using a calibrated standard aneroid or mercury sphygmomanometer or a calibrated standard sphygmomanometer. The change in the MSSBP was calculated comparing the Week 8 readings to the readings taken at Baseline. The change from Baseline in MSSBP was analyzed using an ANCOVA with treatment and country as factors and Baseline MSSBP as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID
Number analyzed (Participants) | 31 | 26 | 31
mmHg | -11.4 (2.96) | -13.1 (3.24) | -12.5 (2.96)

6. Secondary Outcome: Dose/Exposure BP Response Relationship of LCI699, as Measured by Change From Baseline in MSDBP at Week 8
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID
Number analyzed (Participants) | 31 | 26 | 31
mmHg | -4.5 (1.72) | -6.0 (1.88) | -6.1 (1.72)

7. Secondary Outcome: Change From Baseline in Mean 24 Hours, Mean Daytime and Mean Nighttime Systolic Blood Pressure (SBP) at Week 8 LOCF, as Measured by Ambulatory Blood Pressure Measurement (ABPM)
Description: An ABPM measured a participant's blood pressure over a 24-hour period including daytime and nighttime readings, using an automated validated monitoring device from Baseline to Week 8. The 24-hour SBP was calculated by taking the mean of all ambulatory systolic blood pressure readings for the 24-hour period. The change from Baseline in SBP was analyzed using ANCOVA with treatment and country as factors and Baseline MSSBP as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 15 | 19 | 26 | 23 | 23
mmHg
  24-hour Mean SBP | -4.4 (3.22) | -5.7 (2.87) | -6.3 (2.47) | -15.7 (2.59) | -1.0 (2.59)
  Daytime Mean SBP | -4.9 (3.29) | -6.0 (2.92) | -6.3 (2.52) | -15.7 (2.65) | -1.6 (2.65)
  Nighttime Mean SBP | -3.2 (3.49) | -4.8 (3.13) | -7.0 (2.67) | -15.4 (2.81) | 0.4 (2.81)

8. Secondary Outcome: Change From Baseline in Mean 24 Hours, Mean Daytime and Mean Nighttime Diastolic Blood Pressure (DBP) at Week 8 LOCF, as Measured by ABPM
Description: An ABPM measured a participant's blood pressure over a 24-hour period including daytime and nighttime readings, using an automated validated monitoring device from Baseline to Week 8. The 24-hour DBP was calculated by taking the mean of all ambulatory diastolic blood pressure readings for the 24-hour period. The change from Baseline in DBP was analyzed using an ANCOVA with treatment and country as factors and Baseline MSDBP as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 15 | 19 | 26 | 23 | 23
mmHg
  24-hour Mean DBP | 1.0 (2.15) | -3.4 (1.94) | -3.7 (1.67) | -9.6 (1.74) | -0.2 (1.74)
  Daytime Mean DBP | 0.6 (2.31) | -3.6 (2.06) | -3.4 (1.78) | -9.5 (1.86) | -0.8 (1.87)
  Nighttime Mean DBP | 1.9 (2.17) | -2.5 (1.98) | -4.6 (1.69) | -9.6 (1.75) | 1.2 (1.76)

9. Secondary Outcome: Change From Baseline in Mean 24 Hours, Mean Daytime and Mean Nighttime SBP in LCI699 1mg QD Versus LCI699 0.5mg BID Arm at Week 4, as Measured by ABPM
Description: An ABPM measured a participant's blood pressure over a 24-hour period including daytime and nighttime readings using an automated validated monitoring device from Baseline to Week 4. The 24-hour SBP was calculated by taking the mean of all ambulatory systolic blood pressure readings for the 24-hour period. The change from Baseline in SBP was analyzed using an ANCOVA with treatment and country as factors and Baseline MSDBP as a covariate.
Time Frame: Baseline, Week 4
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug. Overall number of participants analyzed signifies the number of participants who were evaluable for this measure. Here, Number Analyzed 'n' represents number of participants who were evaluable for that specific category.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- LCI699 0.5 mg BID: Following a 2-week placebo run-in period, participants received LCI699 0.5 mg, capsules, orally, BID, with or without food for up to 4 weeks.
Arm/Group | LCI699 1 mg QD | LCI699 0.5 mg BID
Number analyzed (Participants) | 18 | 26
mmHg
  24-hour Mean SBP | -7.8 (2.72) | -4.7 (2.29)
  Daytime Mean SBP | -8.1 (2.69) | -5.3 (2.27)
  Nighttime Mean SBP: number analyzed (Participants) | 18 | 25
  Nighttime Mean SBP | -6.8 (3.17) | -4.5 (2.70)

10. Secondary Outcome: Change From Baseline in Mean 24 Hours, Mean Daytime and Mean Nighttime DBP in LCI699 1mg QD Versus LCI699 0.5mg BID Arm at Week 4, as Measured by ABPM
Description: An ABPM measured a participant's blood pressure over a 24-hour period including daytime and nighttime readings using an automated validated monitoring device from Baseline to Week 4. The 24-hour DBP was calculated by taking the mean of all ambulatory diastolic blood pressure readings for the 24-hour period. The change from Baseline in DBP was analyzed using an ANCOVA with treatment and country as factors and Baseline MSDBP as a covariate.
Time Frame: Baseline, Week 4
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | LCI699 1 mg QD | LCI699 0.5 mg BID
Number analyzed (Participants) | 18 | 26
mmHg
  24-hour Mean DBP | -4.3 (1.98) | -2.5 (1.67)
  Daytime Mean DBP | -3.9 (2.04) | -2.6 (1.73)
  Nighttime Mean DBP: number analyzed (Participants) | 18 | 25
  Nighttime Mean DBP | -4.5 (2.21) | -2.8 (1.87)

11. Secondary Outcome: Number of Participants With Adverse Event (AEs), Serious Adverse Events (SAEs), Hyperkalemia, and Hyponatremia
Description: An AE was an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives. SAEs were AEs leading to death, are life-threatening, require hospitalizations or prolongation of hospitalizations, represent an innate malformation or a congenital abnormality. Hyperkalemia was defined as potassium level >5.5 millimoles per liter (mmol/L). It is the medical term that describes a potassium level that's higher than normal. Hyponatremia was defined as sodium level <135 mmol/L. It is the medical term that describes a sodium level that's lesser than normal.
Time Frame: AEs, Hyperkalemia, and Hyponatremia: From start of the study drug treatment up to 10 weeks; SAE: From signing of the informed consent up to 10 weeks
Population: Safety set population included all participants who were randomized and received at least 1 dose of study drug. Here, Number Analyzed represents the number of participants who were evaluable for that specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 32 | 26 | 31 | 33 | 33
Participants
  AE(s) | 15 | 15 | 8 | 13 | 16
  SAE(s) | 0 | 0 | 0 | 1 | 0
  Hyperkalemia [potassium level >5.5 mmol/L]: number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
  Hyperkalemia [potassium level >5.5 mmol/L] | 2 | 0 | 0 | 0 | 1
  Hyperkalemia [potassium level ≥6.0 mmol/L]: number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
  Hyperkalemia [potassium level ≥6.0 mmol/L] | 2 | 0 | 0 | 0 | 0
  Hyponatremia [sodium level <130 and ≥125 mmol/L]: number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
  Hyponatremia [sodium level <130 and ≥125 mmol/L] | 0 | 0 | 0 | 1 | 0
  Hyponatremia [sodium level <135 mmol/L and ≥130mmol/L]: number analyzed (Participants) | 31 | 26 | 31 | 32 | 33
  Hyponatremia [sodium level <135 mmol/L and ≥130mmol/L] | 3 | 2 | 7 | 3 | 2

12. Secondary Outcome: Number of Participants With Cortisol Levels Below 500 Nmol/L at 1 Hour After Adrenocorticotropic Hormone (ACTH) Injection at Week 8
Description: Serum cortisol concentrations at 1 hour after injection were measured to assess the maximum stimulated cortisol level achieved. Potential adrenal suppression was indicated if the serum cortisol concentration was <500 nanomoles per liter (nmol/L) at 1 hour after the injection.
Time Frame: 1-hour post-dose at Week 8
Population: ACTH stimulation test subset population included all participants prior to treatment with LCI699 and at the end of the treatment interval (Week 8).
Measure: Count of Participants; unit: Participants
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
Number analyzed (Participants) | 5 | 4 | 6 | 7 | 7
Participants | 0 | 1 | 4 | 0 | 0

13. Secondary Outcome: Percent Change From Baseline in Renin-Angiotensin-Aldosterone-System (RAAS) Biomarker: Plasma Aldosterone (PA) in LCI699 Compared to Eplerenone 50 mg at Week 8 LOCF
Description: Percent change from Baseline was analyzed by ANCOVA model using PA values measured at Baseline and Week 8 LOCF, with treatment and country as factors and Baseline value as the covariate. Negative percent change from Baseline shows improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change in aldosterone
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID
Number analyzed (Participants) | 27 | 23 | 29 | 31
percent change in aldosterone | -22.3 (0.16) | -30.4 (0.17) | -53.1 (0.15) | 115.0 (0.15)

14. Secondary Outcome: Percent Change From Baseline in RAAS Biomarker: Plasma Renin Activity (PRA) in LCI699 Compared to Eplerenone 50mg at Week 8 LOCF
Description: Percent change from Baseline was analyzed by ANCOVA model using plasma renin values measured at Baseline and Week 8 LOCF, with treatment and country as factors and Baseline value as the covariate. Negative percent change from Baseline shows improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change in PRA
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID
Number analyzed (Participants) | 27 | 20 | 27 | 31
percent change in PRA | 41.6 (0.24) | 74.3 (0.28) | 107.7 (0.24) | 414.1 (0.22)

15. Secondary Outcome: Percent Change From Baseline in RAAS Biomarker: Active Renin (ARC) in LCI699 Compared to Eplerenone 50mg at Week 8 LOCF
Description: Percent change from Baseline was analyzed by ANCOVA model using active renin values measured at Baseline and Week 8 LOCF, with treatment and country as factors and Baseline value as the covariate. Negative percent change from Baseline shows improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change in ARC
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID
Number analyzed (Participants) | 27 | 21 | 28 | 30
percent change in ARC | 73.1 (0.24) | 72.8 (0.27) | 156.4 (0.23) | 430.6 (0.22)

16. Secondary Outcome: Percent Change From Baseline in RAAS Biomarker: Ratio of PA to PRA in LCI699 Compared to Eplerenone 50mg at Week 8 LOCF
Description: Percent change from Baseline was analyzed by ANCOVA model using percent ratio of PA to PRA values measured at Baseline and Week 8 LOCF, with treatment and country as factors and Baseline value as the covariate. Negative percent change from Baseline shows improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change in ratio of PA to PRA
Arm/Group | LCI699 0.25 mg BID | LCI699 1 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID
Number analyzed (Participants) | 26 | 20 | 27 | 31
percent change in ratio of PA to PRA | -46.7 (0.26) | -50.0 (0.29) | -78.3 (0.25) | -57.1 (0.23)

ADVERSE EVENTS:
Time Frame: AEs: From start of the study drug treatment up to 10 weeks; SAE: From signing of the informed consent up to 10 weeks
Description: Safety set population included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- LCI699 1.0 mg QD: Following a 2-week placebo run-in period, participants received LCI699 1 mg, capsules, orally, once daily (QD), with or without food for up to 8 weeks.
Arm/Group | LCI699 0.25 mg BID | LCI699 1.0 mg QD | LCI699 0.5 mg Followed by LCI699 1 mg BID | Eplerenone 50 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/26 | 0/31 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/26 | 0/31 | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 15/32 | 15/26 | 8/31 | 13/33 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCI699 0.25 mg BID (N=32) | LCI699 1.0 mg QD (N=26) | LCI699 0.5 mg Followed by LCI699 1 mg BID (N=31) | Eplerenone 50 mg BID (N=33) | Placebo (N=33)
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCI699 0.25 mg BID (N=32) | LCI699 1.0 mg QD (N=26) | LCI699 0.5 mg Followed by LCI699 1 mg BID (N=31) | Eplerenone 50 mg BID (N=33) | Placebo (N=33)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 3 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Multiple allergies (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood cortisol decreased (Investigations) | 2 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 1 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 4 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.